CLINICAL TRIAL: NCT00429533
Title: A Prospective Randomized Placebo-Controlled Clinical Trial of Dapsone as a Glucocorticoid-Sparing Agent in Maintenance Phase Pemphigus Vulgaris
Brief Title: Efficacy of Dapsone as a Steroid Sparing Agent in Pemphigus Vulgaris
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Jacobus Pharmaceutical (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 51,988
Record Dates: First submitted 2007-01-29; First posted 2007-01-31 (Estimated); Last update posted 2007-02-05 (Estimated); Status verified 2007-02

CONDITIONS: Pemphigus Vulgaris
MeSH Terms: conditions — Pemphigus | interventions — Dapsone

INTERVENTIONS:
Drug: Dapsone

SUMMARY:
The purpose of this 12-month study was to determine the efficacy of dapsone as a glucocorticoid-sparing agent in maintenance phase pemphigus vulgaris.

DETAILED DESCRIPTION:
Patients were entered into the trial on steroids in combination with cytotoxic agents as needed. The steroid dose was the lowest dose at which the patient's disease was controlled before the last flare (see eligibility criteria). The patients were randomized to receive either Dapsone or placebo. Treatment was to be started at a dose of 50 mg and increased by 25 mg increments each week once the hemoglobin was shown not to have dropped by more than 2 gm/dl. The target dose was 150 mg and patients who did not respond could be advanced to 200 mg daily. After beginning treatment, a standardized steroid taper was commenced. A standardized steroid taper was suggested with tapering by 10 mg/wk for doses above 40 mg/day or more slowly if warranted. A slower taper thereafter or an every other day dosing schedule would be elected according to the individual investigator's preference. Flares were treated by increasing the dose of steroids - in the case of a mild flare to the last dose preceding the flare, in the case of a moderate flare by 20 mg/day and in the case of a severe flare by 40 mg/day. Tapering was to be resumed once the disease had stabilized. Disease activity was assessed by a simple scoring system for skin, mucosa, and sites involved. Laboratory assessments initially weekly became monthly once the study medication dosage was stabilized.

ELIGIBILITY:
Inclusion Criteria:

* Histologic evidence compatible with pemphigus vulgaris and direct immunofluorescence evidence of pemphigus vulgaris.
* Chronic disease that has been controlled with steroids and/or cytotoxics, e.g. maintenance phase.
* On prednisone 15 or more mg/day to around 40 mg/day or on prednisone 15 or more mg every other day (qod) to around 40 mg qod.
* Failure to taper steroids below a range of 15 mg/day to around 40 mg/day or 15 mg/qod to around 40 qod without flaring the disease.
* The steroid dosage at which the most recent flare occurred should not be less than 85% of the last (within 30 days) dosage which controlled the disease, i.e. 85% of the baseline steroid dosage. This is to ensure that patients will not have had a recent acute flare at the time of entry into the study, and be in the rapid steroid taper portion of their disease after such a flare.
* Two baseline steroid dosages as determined by prior flares. It is common that patients will be repetitively unable to taper below a certain baseline steroid dose without experiencing a mild flare of their disease. This baseline dose will be determined on two occasions during attempted tapers, and the baseline number then averaged to determine the dose of steroid the patient is on at the time of entry into the study.
* No pulse steroids, pulse cyclosphosphamide, or plasmapheresis within two months of beginning the protocol. This will exclude patients who had recent acute flares of their disease and may be on the rapid steroid taper portion of their disease. The patient must be in maintenance phase, as defined in the criteria listed in e.
* Patient understands the procedures and agrees to participate in the study program by giving written informed consent.

Exclusion Criteria:

* Patients able to taper steroids without recurrence of disease.
* Patients with early, severe disease that have not responded to high doses of prednisone, cytotoxics, plasmapheresis, or other modalities.
* Contraindications to the use of Dapsone, including severe anemia or G6PD deficiency.
* Patient has behavioral problems that might interfere with compliance.
* Pregnancy or breast-feeding.
* Younger than 18 or older than 80 years of age. Since PV is rare in patients younger than 18, it was decided to exclude this potentially different population. It is unlikely that this will exclude many patients. Dapsone induces a hemolytic anemia, which would be a particular problem for patients over age 80, who are more likely to have ischemic heart disease or other atherosclerotic vascular disease.
* History of allergy to dapsone.
* Ischemic heart disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48
Dates: Start 1996-11; Study Completion 2004-02

PRIMARY OUTCOMES:
The ability of patients to taper to ≤7.5mg/day within one year of reaching the maximum dosage of the study drug.

SECONDARY OUTCOMES:
Steroid dosage reduced by more than 25% within 4 months after completing the upward titration of the study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria P. Werth, MD, Study Chair — University of Pennsylvania; Victoria P. Werth, MD, Principal Investigator — University of Pennsylvania; Diana Chen, MD, Principal Investigator — Northwestern University; Warren R Heymann, MD, Principal Investigator — Cooper Hospital/University Medical Center; Neil Korman, MD, Principal Investigator — Case Western Reserve University School of Medicine; Amit Pandya, MD, Principal Investigator — University of Texas; M J Rico, MD, Principal Investigator — The New York VA Medical Center - New York University; Michael D Tharp, MD, Principal Investigator — Rush University Medical Center
Locations (8):
- United States (8):
  - Northwestern University Medical Center, Chicago, Illinois
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - Henry Ford Hospital, Detroit, Michigan
  - Cooper Hospital/University Medical Center, Camden, New Jersey
  - The New York VA Medical Center, New York University, New York, New York
  - Case Western Reserve University School of Medicine, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas, Dallas, Texas

REFERENCES:
- [Derived] Werth VP, Fivenson D, Pandya AG, Chen D, Rico MJ, Albrecht J, Jacobus D. Multicenter randomized, double-blind, placebo-controlled, clinical trial of dapsone as a glucocorticoid-sparing agent in maintenance-phase pemphigus vulgaris. Arch Dermatol. 2008 Jan;144(1):25-32. doi: 10.1001/archderm.144.1.25. PMID 18209165